CLINICAL TRIAL: NCT03000179
Title: Pilot Study to Investigate the Safety and Efficacy of Avelumab Monotherapy in Patients With Advanced or Metastatic Adenocarcinoma of the Small Intestine
Brief Title: Safety and Efficacy of Avelumab in Small Intestinal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); EMD Serono (Industry)
Responsible Party: Principal Investigator, Dana Cardin, MD, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 1679
Record Dates: First submitted 2016-12-06; First posted 2016-12-21 (Estimated); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Adenocarcinoma
Keywords: small bowel cancer, small bowel carcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab Monotherapy (Experimental): Participants receive avelumab by IV infusion following pretreatment with H1 blockers and acetaminophen once every 2 weeks.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab through a vein once every 2 weeks

SUMMARY:
This is a single-agent, open label, one-arm phase 2 pilot study of avelumab in patients with advanced or metastatic adenocarcinoma of the small intestine.

DETAILED DESCRIPTION:
Primary Objectives

* To describe any antitumor activity of avelumab monotherapy, as measured by the response rate in patients with advanced or metastatic small intestinal adenocarcinoma.
* To describe the safety profile of avelumab monotherapy in patients with advanced or metastatic small intestinal adenocarcinoma.

Secondary Objectives

* To determine overall survival, progression-free survival, and duration of response of avelumab monotherapy in patients with advanced small intestinal adenocarcinoma.
* To evaluate the association of tumor PD-L1 and PD-1 expression, MSI status, lymphocytic infiltration, and somatic mutation burden with response.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent.
* Male or female ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Histologically confirmed adenocarcinoma of the small intestine that is advanced (not amenable to surgery) or metastatic (clinical stage IV). For the purposes of this study, ampullary tumors are considered a part of the duodenum and are classified as adenocarcinomas of the small intestine.
* At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria that has not been previously irradiated and which can be followed by CT or MRI.
* Adequate organ function including:

  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  * Platelets ≥ 100 × 109/L
  * Hemoglobin ≥ 9/g/dL (may have been transfused)
  * Total serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 × ULN (or ≤ 5 × ULN if liver metastases are present)
  * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 30 mL/min as calculated using the Cockcroft-Gault (CG) equation
* Archival tissue [paraffin block(s) or unstained slides from paraffin block(s)] from the primary tumor and/or a metastatic site judged reasonably available prior to initiating treatment, or willingness to undergo fresh pre-treatment tumor biopsy. (Prior to initiating treatment, the screening team must have documentation that an archival or fresh tumor specimen has been requested from a local or outside facility. However, physical possession of requested tissue or waiting for histological analysis or confirmation that an acquired specimen contains tumor tissue sufficient for analysis is not a requirement prior to initiating treatment.) If no archival tissue is available and patient consents to a fresh biopsy, but the patient's lesion is deemed inaccessible to safe biopsy, the patient will be allowed to enroll if otherwise eligible.
* Female patients of childbearing potential and male patients able to father children who have female partners of childbearing potential must agree to use one highly effective method (defined as less than 1% failure rate per year) and one additional effective method of contraception (Appendix 4) from 15 days prior to first trial treatment administration until at least 60 days after study participant's final dose of avelumab.

  * Females of childbearing potential are defined as those who are not surgically sterile or post-menopausal (i.e. patient has not had a bilateral tubal ligation, a bilateral oophorectomy, or a complete hysterectomy; or has not been amenorrheic for 12 months without an alternative medical cause). Post-menopausal status in females under 55 years of age should be confirmed with a serum follicle-stimulating hormone (FSH) level within laboratory reference range for postmenopausal women.
  * Male patients able to father children are defined as those who are not surgically sterile (i.e. patient has not had a vasectomy).
* Serum pregnancy test (for females of childbearing potential) negative at screening.
* Re-enrollment of a subject that has discontinued the study as a pre-treatment screen failure (i.e. a consented patient who did not receive avelumab) is permitted. If re-enrolled, the subject must be re-consented. Only the screening procedures performed outside of protocol-specified timing must be repeated.

Exclusion Criteria:

* There is no restriction on the number of prior therapies. However, prior therapy with antibody or drug specifically targeting T cell regulatory proteins, including but not limited to the following is not allowed: Prior immunotherapy with IL-2 or IFN-α, or an anti-PD-1 (including nivolumab), anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyteassociated antigen-4 (CTLA-4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Within 28 days before first dose of avelumab: Anti-cancer treatment, major surgery requiring general anesthesia, or the use of any investigational agent.
* Within 14 days before first dose of avelumab: Therapeutic or palliative radiation therapy. (Subjects receiving bisphosphonate or denosumab are eligible provided treatment was initiated at least 14 days before the first dose of avelumab.)
* Current use of immunosuppressive medication, except the following:

  * Subjects are permitted the use of corticosteroids with minimal systemic absorption (e.g. topical, ocular, intra-articular, intranasal, and inhaled);
  * Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent are permitted;
  * A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g. CT scan premedication against contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by a contact allergen) is permitted.
* Previous malignant disease other than adenocarcinoma of the small intestine within the last 5 years, with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ considered curatively treated (i.e. complete remission achieved at least 2 years prior to first dose of avelumab AND additional therapy not required while receiving study treatment).
* All subjects with brain metastases, expect those meeting the following criteria:

  * Brain metastases that have been treated locally and are clinically stable for at least 2 weeks prior to enrollment
  * No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable.
  * Subjects must be either off steroids or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent)
* Receipt of any organ transplantation including allogeneic stem-cell transplantation.
* Significant acute or chronic infections requiring systemic therapy.

  * Known history of testing positive for human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS).
  * Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
* Active autoimmune disease with reasonable possibility of clinically significant deterioration when receiving an immunostimulatory agent:

  * Subjects with Type 1 diabetes mellitus, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
* Interstitial lung disease that is symptomatic or which may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Uncontrolled asthma [defined as having 3 or more of the following features of partially controlled asthma within 28 days prior to starting study treatment: Daytime symptoms more than twice per week, any limitation of activities, any nocturnal symptoms/awaking, need for reliever/rescue inhaler more than twice per week, or known lung function (PEF or FEV1) without administration of a bronchodilator that is < 80% predicted or personal best (if known)].
* Current symptomatic congestive heart failure (New York Heart Association > class II), unstable cardiac arrhythmia requiring therapy (e.g. medication or pacemaker), unstable angina (e.g. new, worsening or persistent chest discomfort), or uncontrolled hypertension (systolic > 160 mmHg or diastolic > 100mmHg). Or any of the following occurring within 6 months (180 days) prior to first dose of avelumab: Myocardial infarction, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack, or serious cardiac arrhythmia requiring medication. (Use of antihypertensive medication to control blood pressure is allowed.)
* Concurrent treatment with a non-permitted drug.
* Requirement of anticoagulant therapy with oral vitamin K antagonists such as Coumadin (warfarin). Low-dose anticoagulants for the maintenance of patency in a central venous access device or the prevention of deep vein thrombosis or pulmonary embolism is allowed. Therapeutic use of low molecular weight heparin is allowed.
* Persisting toxicity related to prior therapy that has not reduced to Grade 1 [National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.03; however, alopecia and sensory neuropathy Grade ≤ 2 is acceptable.
* Known severe (Grade ≥ 3 NCI-CTCAE v4.03) hypersensitivity reactions to monoclonal antibodies, including hypersensitivity to the investigational agent or any component in its formulations, or history of anaphylaxis.
* Vaccination within 28 days of the first dose of avelumab and while on trial is prohibited, except for administration of inactivated vaccines (for example, inactivated influenza vaccine).
* Pregnant or breastfeeding females.
* Known alcohol or drug abuse.
* Prisoners or subjects who are involuntarily incarcerated.
* Other severe acute or chronic medical condition, including colitis, inflammatory bowl disease, pneumonitis, pulmonary fibrosis, or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Cardin, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled onto this study at Vanderbilt University Medical Center in Nashville, TN from March 2017 to August 2019. The study closed early due to low accrual.
Period: Overall Study
Arm/Group | Avelumab Monotherapy
Started | 8
Completed | 6
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab Monotherapy
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate as Measured Using RECIST 1.1
Description: Response rate is the proportion of patients with overall complete (CR) or partial response(PR) among patients with valuable response outcome. Overall response will consider both target and non-target lesions, as well as new lesions.
  Target lesions by CT/MRI: CR: Disappearance of all target lesions. PR: >= 30% decrease in the sum of diameters of target lesions. Progressive Disease (PD): >= 20% increase in the sum of diameters of target lesions, In addition, the sum must also demonstrate an absolute increase of at least 5 mm or appearance of new lesions. Non-target lesions: CR: Disappearance of all target lesions. Non-CR/Non-PD: Persistence of one or more non-target lesion(s) and/or maintenance of applicable tumor marker level above the normal limits. PD: progression of existing non-target lesions.
Time Frame: Measured every 8 weeks through study completion, an average of 1 year
Population: Patients with advanced small intestinal adenocarcinoma or ampullary tumors, efficacy-evaluable.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Avelumab Monotherapy
Number analyzed (Participants) | 7
proportion of participants | 0.29 [0.08 to 0.64]

2. Primary Outcome: Number of Patients With Each Worst-Grade Toxicity
Description: To describe the safety profile of avelumab monotherapy in patients with advanced or metastatic small intestinal adenocarcinoma
Time Frame: On-study date to 30 days following final dose of study drug, or until the event is resolved, stabilized, or determined to be irreversible by the participating investigator if beyond 30 days.
Population: all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab Monotherapy
Number analyzed (Participants) | 8
Participants
  Anemia, Grade 1 | 2
  Fatigue, Grade2 | 1
  Infusion related reaction. Grade2 | 2
  Alanine aminotransferase increased, Grade 1 | 1
  Alkaline phosphatase increased, Grade 1 | 1
  Anorexia, Grade 2 | 1
  Blood bilirubin increased, Grade1 | 1
  Diarrhea, Grade 1 | 1
  Diabetic ketoacidosis, Grade 4 | 1
  Back pain, Grade 1 | 1
  Diverticulitis per upper GI series, Grade 2 | 1
  Hypokalemia, Grade 3 | 1
  Hyponatremia, Grade 3 | 1
  Nausea, Grade 2 | 1
  Rash maculo-papular, Grade 1 | 1
  Urticaria, Grade 1 | 1

3. Secondary Outcome: Overall Survival
Description: On study date until death from any cause
Time Frame: Every 3 months after completing treatment up to 5 years
Population: all participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Monotherapy
Number analyzed (Participants) | 8
months | 6.4 [3.8 to NA] — Insufficient number of patients with the death event

4. Secondary Outcome: Progression Free Survival
Description: On-study date until disease progression or death. Progression is >= 20% increase in the sum of diameters of target lesions or non-target lesions, or appearance of new lesions.
Time Frame: On-study date to lesser of date of progression or date of death from any cause measured up to 3 years after treatment
Population: all participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab Monotherapy
Number analyzed (Participants) | 8
months | 3.4 [3.0 to NA] — Insufficient number of patients with progression.

5. Secondary Outcome: Duration of Response
Description: Time from tumor response date to disease progression or death for any reason.
Time Frame: Date of first partial or complete response as defined by RECIST 1.1 criteria to date of recurrence or disease progression up to 3 years
Population: Patients who had partial response.
Measure: Median (Full Range); unit: months
Arm/Group | Avelumab Monotherapy
Number analyzed (Participants) | 2
months | 10.9 [3.0 to 18.8]

ADVERSE EVENTS:
Time Frame: From study entry to up to 28 days from the last dose of avelumab up to approximately 1 year.
Arm/Group | Avelumab Monotherapy
All-Cause Mortality (participants affected / at risk) | 6/8
Serious Adverse Events (participants affected / at risk) | 7/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab Monotherapy (N=8)
Diabetic Ketoacidos (Endocrine disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Bacteremia bloodstream infection (Infections and infestations) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Sepsis (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab Monotherapy (N=8)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 4 (6)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (20)
Lymphocyte count decreased (Investigations) | 4 (8)
Alkaline phosphatase increased (Investigations) | 3 (8)
Weight loss (Investigations) | 3 (5)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (2)
INR increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 2 (4)
Chills (General disorders) | 1 (1)
Limb edema (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (8)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Investigations) | 2 (7)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Small intestine infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Syncope (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
memory impairement (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Couph (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Thromboembolic event (Nervous system disorders) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Generalized muscle weaknes (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Extremity pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Psychosis (Psychiatric disorders) | 1 (2)
Restlessness (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03000179/Prot_SAP_000.pdf